CLINICAL TRIAL: NCT05116098
Title: Randomized Clinical Trial: IS Zinc and Zinc Ionophere EGCG as Supplement Improve Outcome of Active Pulmonary Tuberculosis
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ministry of Health, Saudi Arabia (Other Government)
Responsible Party: Principal Investigator, Amr kamel khalil Ahmed, Ministry of Health, Saudi Arabia, Ministry of Health, Saudi Arabia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: tuberculosis treatment
Record Dates: First submitted 2021-10-20; First posted 2021-11-10 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-11

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis | interventions — Zinc; epigallocatechin gallate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- 100 pulmonary positive patients on tb protocol adding to supplement zinc 50 mg 400 mg once daily (Active Comparator)
  Interventions: Combination Product: zinc 50 mg + Epigallocatechin gallate
- control group 100 patients only on tuberculosis national protocol (Placebo Comparator)
  Interventions: Combination Product: zinc 50 mg + Epigallocatechin gallate

INTERVENTIONS:
Combination Product: zinc 50 mg + Epigallocatechin gallate — ZINC 50 MG and EGCG 200mg oral daily for 1 month

SUMMARY:
Tuberculosis is still global burden disease at all the word and effect on quality life of patients and affect on health authorities because the cost of medicine and health cost .

* A total of 1.4 million people died from TB in 2019 (including 208 000 people with HIV). Worldwide, TB is one of the top 10 causes of death and the leading cause from a single infectious agent (above HIV/AIDS).
* In 2019, an estimated 10 million people fell ill with tuberculosis (TB) worldwide. 5.6 million men, 3.2 million women and 1.2 million children. TB is present in all countries and age groups. But TB is curable and preventable.
* In 2019, 1.2 million children fell ill with TB globally. Child and adolescent TB is often overlooked by health providers and can be difficult to diagnose and treat.
* In 2019, the 30 high TB burden countries accounted for 87% of new TB cases. Eight countries account for two thirds of the total, with India leading the count, followed by Indonesia, China, the Philippines, Pakistan, Nigeria, Bangladesh and South Africa. ( WHO) All TB cases and 92.5% controls were zinc deficient. The odds of TB cases with deficiencies of vitamin A and zinc was 2.3 (95% CI: 1.1 to 4.8) times more likely as compared to the controls. More than 80% of all participants had below average fulfilment of energy and vitamin A intakes. (7) Zinc is necessary for intact immune health and defense against infection but there are common health problem deficiency at developing countries and so zinc needs as supplement and the second problem zinc need helper for transfer through plasma membrane so zinc ionophore is a best solution as this problem so the investigators can use zinc ionophore as helper for zinc to enter the cells for autophagy

DETAILED DESCRIPTION:
M. tuberculosis -infected PMs, in vitro, elaborated IL-6 as the only major cytokine, which was significantly inhibited by anti-TB drugs. Therefore, IL-6 can be developed as a potential biomarker or biosignature to assess the success of the treatment of TB. (1) Tuberculosis is a global health problem, and there is even an increase in cases of multidrug-resistant tuberculosis in the world. Therefore, research is needed that can find new anti-tuberculosis drugs (OAT) that are more effective for tuberculosis treatment. In this study, the effect of (-)-epigallocatechin-gallate (EGCG) of tea leaves (Camellia sinensis) combined with the first-line OAT will be observed, in order to find out whether EGCG has anti-tuberculosis activity and can increase the potential of first-line OAT in-vitro. The anti-tuberculosis activity of EGCG was determined by broth dilution method using Middlebrook 7H9 media at concentration of 50, 100, 150, dan 200 ppm, then the potential of first-line OAT before and after combined with the EGCG was observed. The results showed that the activity of EGCG at concentration 50 ppm and 100 ppm could inhibit the Mycobacterium tuberculosis growth by 80%, at concentration 150 ppm by 90%, and at concentration 200 ppm by 100%. First-line OAT activity before combined with EGCG was ≥ 90% at 5 ppm rifampicin, 0.5 ppm isoniazid, 50 ppm pyrazinamide, and 5 ppm ethambutol. Whereas after combined with EGCG, the potential of each drug increased, marked by anti-tuberculosis activity achieved ≥ 90% at lower concentrations, i.e. rifampicin 0.5 ppm, isoniazid 0.25 ppm, pyrazinamide 20 ppm, and ethambutol 2 ppm. These results indicated that the potential of each first-line OAT increases after being combined with EGCG, and EGCG has potentiation effect when combined with those drugs. In conclusion, EGCG can increase the first-line OAT activity (2)

The down-regulation of TACO gene expression by epigallocatechin-3-gallate was accompanied by inhibition of mycobacterium survival within macrophages as assessed through flow cytometry and colony counts. Based on these results, the investigators propose that epigallocatechin-3-gallate may be of importance in the prevention of tuberculosis infection. (3) The effectiveness of anti-tuberculosis treatment was improved during the first two months by vitamin A and zinc supplementation," Dr. Clive E. West, a professor in the department of nutrition at Wageningen University in the Netherlands, and colleagues write in the April issue of the American Journal of Clinical Nutrition (2002;75:720-727). Previous research has shown that TB patients often suffer from malnutrition, which can weaken immune response and increase disease susceptibility. The addition of vitamin A and zinc has been observed to boost the immune response in these patients. Patients who received the supplements were twice as likely to have eliminated the TB bacteria from the mucus coughed up from their lungs by two weeks than the group receiving only standard drug treatment, and maintained that difference for seven weeks. These patients also had a greater reduction in abnormalities or lesions on their chest x-rays than those not taking the supplements. Reducing the amount of potentially contagious bacteria present in patients' sputum would cut the rate at which they spread TB to others, the researchers noted. (4) The effect of green tea extract supplementation on sputum smear conversion and weight changes in pulmonary TB patients: A randomized controlled trial (5) Zinc is an essential micronutrient (34, 40-42), and its tissue and plasma levels are influenced by dietary intake (38, 42). While severe zinc deficiency is rare in the developed world, moderate zinc deficiency is widespread, concentrated in elderly populations (42-45), and can be exacerbated in critically ill patients (33, 46-49). the investigators demonstrate that both genetic MT deficiency and dietary zinc deficiency potentiate lung injury in mechanically ventilated mice, consistent with an essential role for the zinc/MT system in protecting the lung from injurious stretch. To demonstrate clinical relevance of our findings, the investigators show that humans who go on to develop ARDS exhibit lower plasma zinc levels. Taken together, our results suggest that failure of essential stretch-adaptive responses, in this case associated with a remediable dietary deficiency among hospitalized patients, may play an important role in injury responses propagated by MV. (6)

ELIGIBILITY:
Inclusion Criteria:

1. new diagnosed pulmonary positive t.b patients
2. age above 18 years
3. any patients with HIV and immuncromoised with t.b patients
4. patients with covid 19 and t.b
5. patients with drug t.b resistant
6. male or female
7. all races African or Asian or white -

Exclusion Criteria:

1- less than 18 years 2- pregnant female 3- on another supplement

-

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-11-30 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
sputum analysis at start of treatment and after one month | 6 month
  percentage of conversion sputum samples converted from positive to negative after one month

SECONDARY OUTCOMES:
measurement of serum or plasma zinc at all participants | 6 month
measurement of serum interleukin 6 | 6 month
  measurement of serum interleukin 6
serum Adenosine deaminase (ADA) | 6 month
  measurement of serum Adenosine deaminase (ADA)

IPD SHARING:
Plan to Share IPD: Undecided